CLINICAL TRIAL: NCT03462758
Title: Early vs. Interval Postpartum IUD Insertion: A Multi-site Randomized Controlled Trial
Brief Title: Early vs. Interval Postpartum IUD Insertion
Acronym: EPPIUD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of New Mexico (Other); United States Naval Medical Center, San Diego (U.S. Federal Agency); University of Illinois at Chicago (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, Sarah Averbach, MD MAS, Associate Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 172101
Record Dates: First submitted 2018-01-24; First posted 2018-03-13 (Actual); Results first posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Contraception
Keywords: Mirena; ParaGard; Skyla; Liletta; Kyleena; Intrauterine Device; Intrauterine System; Postpartum; Expulsion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Control Group (Other): IUD placed 6-8 weeks postpartum (standard of care, interval placement)
  Interventions: Device: IUD
- Intervention Group (Experimental): IUD placed 2-4 weeks postpartum (early postpartum placement, EPP)
  Interventions: Device: IUD

INTERVENTIONS:
Device: IUD — Postpartum IUD placement
  Other Names: Mirena, Kyleena, Skyla, Liletta, ParaGard

SUMMARY:
Intrauterine devices (IUDs) are historically placed at a six-week postpartum visit for women who desire intrauterine contraception after delivery. A two-week postpartum visit could be a convenient time for women to receive contraception, including IUDs. Offering women IUDs at two-weeks postpartum may decrease the risk of undesired pregnancy and rapid repeat pregnancy. This study will compare IUD insertion at two different times after delivery: two-weeks and six-weeks postpartum. This will allow researchers to assess whether the timing of IUD placement affects whether an IUD is expelled, or pushed out of it's ideal location.

DETAILED DESCRIPTION:
The purpose of this study is to determine the proportion of IUDs inserted in the Early Postpartum (EPP) period that are expelled at 6 months postpartum. This prospective, multi-site randomized trial will enroll approximately 404 women at three large academic hospitals in the United States.

Women will be recruited who are interested in receiving a levonorgestrel-IUD or a copper-IUD after delivery. Postpartum women who desire an IUD will be randomized to EPP IUD insertion (between 14-28 days PP) or interval postpartum IUD insertion (42-56 days PP) and the proportion of IUDs expelled will be compared between groups at 6 months postpartum. All women will be seen in clinic at 6-8 weeks and 6 months postpartum. Women randomized to EPP IUD placement will be seen at 2-3 weeks postpartum.

Provider perspectives of EPP IUD placement will also be evaluated, as will whether these attitudes change after 6 to 9 months of providing early postpartum IUDs.

ELIGIBILITY:
Inclusion Criteria:

* Gave birth less than or equal to 10 days ago
* Desires to use an IUD for Contraception (either copper or levonorgestrel)
* Willing and able to sign an informed consent
* Willing to comply with the study protocol
* Age greater than or equal to 18 years
* English or Spanish speaking

Exclusion Criteria:

* Uterine anomaly or leiomyomata which would not allow placement of an IUD
* Desire for repeat pregnancy in less than 6 months
* Evidence of intrauterine infection (chorioamnionitis or postpartum endometritis) treated with antibiotics
* Ruptured uterus at the time of delivery
* Received a postpartum tubal ligation or immediate postpartum IUD or implant at delivery
* Incarcerated women or women with significant cognitive impairment
* 4th degree perineal laceration sustained at delivery
* Any medical contraindication to IUD per the US Centers for Disease Control (CDC) Medical Eligibility Criteria
* Suspicion for new pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2018-03-20 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Averbach, MD, MAS, Principal Investigator — University of California, San Diego
Locations (4):
- United States (4):
  - University of California, San Diego, La Jolla, California
  - Naval Medical Center San Diego, San Diego, California
  - University of Illinois at Chicago, Chicago, Illinois
  - University of New Mexico, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berkley HH, Lutgendorf MA, Kully G, Raiciulescu S, Stortz SK, Hinz E, Hofler LG, Averbach S. Pain With Early Postpartum Intrauterine Device Placement. O G Open. 2025 Jun 12;2(3):e088. doi: 10.1097/og9.0000000000000088. eCollection 2025 Jun. PMID 41000085
- [Derived] Averbach S, Kully G, Hinz E, Dey A, Berkley H, Hildebrand M, Vaida F, Haider S, Hofler LG. Early vs Interval Postpartum Intrauterine Device Placement: A Randomized Clinical Trial. JAMA. 2023 Mar 21;329(11):910-917. doi: 10.1001/jama.2023.1936. PMID 36943214

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from inpatient postpartum hospital units of the study sites. The first participant was enrolled on March 26, 2018 and the final participant was enrolled on July 29, 2021.
Pre-assignment Details: 404 patients enrolled in the study, all of whom met inclusion criteria.
Groups:
- Interval Postpartum IUD Placement: IUD placed 6-8 weeks postpartum (standard of care, interval placement)
  IUD: Postpartum IUD placement
- Early Postpartum IUD Placement: IUD placed 2-4 weeks postpartum (early postpartum placement, EPP)
  IUD: Postpartum IUD placement
Period: Overall Study
Arm/Group | Interval Postpartum IUD Placement | Early Postpartum IUD Placement
Started | 201 | 203
Completed | 145 | 149
Not Completed | 56 | 54
Not completed — Chose no or other method of contraception | 20 | 23
Not completed — Lost to follow-up before IUD placement | 14 | 12
Not completed — Unsuccessful IUD placement attempt | 3 | 3
Not completed — Medical contraindication | 2 | 2
Not completed — Lost to follow-up after IUD placement | 17 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interval Postpartum IUD Placement | Early Postpartum IUD Placement | Total
Number analyzed (Participants) | 201 | 203 | 404
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.0 (5.5) | 29.8 (5.2) | 29.9 (5.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 201 | 203 | 404
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 93 | 82 | 175
  Not Hispanic or Latino | 108 | 121 | 229
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 6 | 9
  Asian | 12 | 10 | 22
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 2
  Black or African American | 20 | 26 | 46
  White | 114 | 114 | 228
  More than one race | 48 | 42 | 90
  Unknown or Not Reported | 4 | 3 | 7
Education [Count of Participants; unit: Participants]
  High school degree or less | 122 | 111 | 233
  College degree | 38 | 43 | 81
  Graduate degree | 41 | 49 | 90
Employment [Count of Participants; unit: Participants]
  Full time | 92 | 100 | 192
  Unemployed/Retired | 69 | 66 | 135
  Part time | 24 | 22 | 46
  Student | 16 | 15 | 31
Type of most recent delivery [Count of Participants; unit: Participants]
  Vaginal | 152 | 155 | 307
  Cesarean | 49 | 48 | 97
Parity [Count of Participants; unit: Participants]
  Multiparous | 130 | 135 | 265
  Primiparous | 71 | 68 | 139
Type of IUD [Count of Participants; unit: Participants] — Population: All participants who had an IUD placed at any time between randomization and 6-month follow-up.
  Participants
    number analyzed (Participants) | 162 | 163 | 325
    52-mg levonorgestrel | 111 | 101 | 212
    Copper | 49 | 56 | 105
    19.5-mg/13.5-mg levonorgestrel | 2 | 6 | 8
Ultrasonography used [Count of Participants; unit: Participants] — Population: All participants who had an IUD placed at any time between randomization and 6-month follow-up.
  Participants
    number analyzed (Participants) | 162 | 163 | 325
    During placement | 4 | 31 | 35
    After placement only | 5 | 4 | 9
    None | 153 | 128 | 281
Lactating at time of IUD insertion [Count of Participants; unit: Participants] — Population: Excluding missing values on lactation status.
  Participants
    number analyzed (Participants) | 151 | 156 | 307
    Yes | 127 | 139 | 266
    No | 24 | 17 | 41
Clinician performing IUD insertion [Count of Participants; unit: Participants] — Population: Excluding missing values on clinician type.
  Participants
    number analyzed (Participants) | 157 | 162 | 319
    Faculty physician | 75 | 93 | 168
    Advanced practice clinician | 50 | 51 | 101
    Resident physician | 32 | 18 | 50

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With an IUD Expulsion (Complete) at 6 Months
Description: Complete IUD expulsion will be defined as an IUD which no longer in the uterus on speculum exam and transvaginal ultrasound will be performed on all patients at 6 months postpartum to confirm IUD use
Time Frame: 6 months postpartum
Population: Modified intention to treat (MITT) analysis: those who received an IUD within 6 months of delivery whose outcome was known at the end of the study period.
Measure: Count of Participants; unit: Participants
Arm/Group | Interval Postpartum IUD Placement | Early Postpartum IUD Placement
Number analyzed (Participants) | 145 | 149
Participants | 0 | 3

2. Secondary Outcome: Proportion of Participants Using an IUD at 6 Months
Description: IUD utilization will be defined as intrauterine use of an IUD at 6 months postpartum. A speculum exam and transvaginal ultrasound will be performed on all patients at 6 months postpartum to confirm IUD use
Time Frame: 6 months postpartum
Population: Percentages based on total study sample rather than MITT analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Interval Postpartum IUD Placement | Early Postpartum IUD Placement
Number analyzed (Participants) | 201 | 203
Participants | 139 | 141

3. Secondary Outcome: Proportion of Participants With an IUD Expulsion (Partial) at 6 Months
Description: Partial IUD expulsions will be diagnosed in any participant found to have an IUD in which part of the body of the IUD is noted to be coming through the external cervical os on speculum exam.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Interval Postpartum IUD Placement | Early Postpartum IUD Placement
Number analyzed (Participants) | 145 | 149
Participants | 11 | 14

4. Secondary Outcome: Proportion of Participants With a Pelvic Infection Within 6 Months
Description: Pelvic infection requiring antibiotics will be ascertained by patient report and/or medical record review.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Interval Postpartum IUD Placement | Early Postpartum IUD Placement
Number analyzed (Participants) | 145 | 149
Participants | 0 | 3

5. Secondary Outcome: Patient Satisfaction With IUD Assessed on a Five-point "Likert" Scale for Satisfaction, an Ordinal Scale That Measure Levels of Agreement/Disagreement
Description: Participants are asked how much they agree with the statement "I am satisfied with using this IUD." Answers are valued 1-5, with 1 Strongly Agree, 2 Agree, 3 Neutral, 4 Disagree, and 5 Strongly Disagree. 1=Strongly Agree is considered the best outcome, 5=Strongly disagree is considered the worst outcome. Outcome reported is those who were very satisfied or satisfied.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Interval Postpartum IUD Placement | Early Postpartum IUD Placement
Number analyzed (Participants) | 145 | 149
Participants | 116 | 129

6. Secondary Outcome: Proportion of Participants With an IUD Perforation at 6 Months
Description: IUD perforations through the uterus will be diagnosed when an IUD visible is not visible on transvaginal ultrasound of the uterus but is visible on x-ray of the abdomen or pelvis.
Time Frame: 6 months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Interval Postpartum IUD Placement | Early Postpartum IUD Placement
Number analyzed (Participants) | 145 | 149
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Interval Postpartum IUD Placement | Early Postpartum IUD Placement
All-Cause Mortality (participants affected / at risk) | 0/145 | 0/149
Serious Adverse Events (participants affected / at risk) | 0/145 | 0/149
Other Adverse Events (participants affected / at risk) | 0/145 | 0/149

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT03462758/Prot_SAP_000.pdf